CLINICAL TRIAL: NCT05329792
Title: A Phase II Study of L19IL2/L19TNF in Patients With Skin Cancers Amenable to Intralesional Treatment
Brief Title: L19IL2/L19TNF in Skin Cancer Patients
Acronym: IntriNSiC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2TNFBASK-04/21
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: BCC - Basal Cell Carcinoma; SCC - Squamous Cell Carcinoma; Merkel Cell Carcinoma; Keratoacanthoma of Skin; Malignant Adnexal Tumors of the Skin (MATS); Tumors From Cutaneous T-cell Lymphoma (CTCL); Kaposi Sarcoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Carcinoma, Merkel Cell; Sarcoma, Kaposi | interventions — daromun

STUDY DESIGN:
Intervention Model Description: Phase II, open label, multicentric, proof-of-principle basket trial in patients with malignant tumors of the skin amenable to intratumoral injection, and in a curative or neoadjuvant or palliative intention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm with L19IL2 /L19TNF (Experimental): 70 patients will be enrolled and treated with a mixture of L19IL2 and L19TNF once weekly for 4 consecutive weeks. The total dose/volume will be distributed among the target lesions defined at screening via single or multiple intralesional injections, according to lesions' size and number.
  Interventions: Drug: L19IL2/L19TNF

INTERVENTIONS:
Drug: L19IL2/L19TNF — Patients will be treated with a mixture of L19IL2 and L19TNF once weekly for 4 consecutive weeks
  Other Names: bifikafusp alfa/onfekafusp alfa

SUMMARY:
Phase II, open label, multicentric, proof-of-principle basket trial in patients with malignant tumors of the skin amenable to intratumoral injection, and in a curative or neoadjuvant or palliative intention.

DETAILED DESCRIPTION:
Phase II, open label, multicentric, proof-of-principle basket trial in patients with malignant tumors of the skin amenable to intratumoral injection, and in a curative or neoadjuvant or palliative intention.

In the study, 70 patients will be enrolled and treated with a mixture of L19IL2 and L19TNF once weekly for 4 consecutive weeks. The total dose/volume will be distributed among the target lesions defined at screening via single or multiple intralesional injections, according to lesions' size and number.

Tumor assessment:

* Tumor assessment (TA) visits will be performed at Week 12 (Day 78 from the beginning of treatment), then every 8 weeks and up to Week 52 after beginning of treatment. For confirmation of objective responses, unscheduled visits will be performed 4 weeks after the visit, which the objective response was first recorded at.
* During each TA visit, measurement of tumor lesions and documentation (photographic documentation with use of a caliper for cutaneous lesions; ultrasound for subcutaneous lesions; imaging techniques as deemed appropriate/necessary by treating physician) will be performed. The choice of the most suitable instrumental technique to measure and document evolution of the disease will be made by the treating physician at baseline screening, the same technique will have to be used for all following tumor assessments.
* Histological assessment of tumor tissue: estimation of percent of residual viable tumor cells and tumor infiltration with immune responsive cell. Locally performed histological specimen assessment will be centrally reviewed.

After confirmed partial responses, surgery with curative intent is allowed (if considered feasible and of potential benefit for the patients by the treating physician) and will be performed no later than 4 weeks after the TA visit at which the partial response is confirmed.

Safety assessment:

• The safety profile of intratumoral administration of L19IL2/L19TNF will be assessed throughout the study. A complete safety assessment will be performed at the safety visit.

Human-anti-fusion protein antibodies (HAFA) assessment:

• The possible development of antibodies against L19IL2 or L19TNF will be verified. Samples will be collected before L19IL2/L19TNF administration at Days 1, 22 and Day 78 (TA visit).

A Data and Safety Monitoring Board (DSMB), composed of expert dermato-oncologists, will evaluate safety and efficacy data after the first 20 patients and will formulate recommendations for the prosecution of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient participation to the present study is subjected to the positive evaluation of a local interdisciplinary tumor board, in the context of available treatment alternatives. Whatever the tumor (list of eligible tumors below) the local interdisciplinary tumor board has to consider that a local response to injection of L19IL2/L19TNF may be of benefit for the patient, in the context of this tumor and available therapeutic opportunities, benefit defined by any of the following objectives: (1) to avoid surgery considered difficult or mutilating or (2) as a neoadjuvant treatment with the objective to permit surgery considered initially impossible, or to facilitate surgery considered difficult or mutilating, or to secure surgery considered of uncertain effect or (3) as a salvage treatment to control a tumor proved resistant to treatment alternatives or (4) as a palliative treatment improving patient comfort.
2. Patient must have at least one skin tumor that is amenable to intratumoral injection.
3. All tumors must be histologically confirmed before treatment.
4. Patients with skin tumors eligible to the present study include:

   * BCC patients with difficult-to-treat lesions: as defined by EADO operational staging system (stages IIa to IIIb) [1]. Patients must either (i) have already received, or (ii) have progressed after, or (iii) be resistant to, or (iv) not be candidate to all possible alternative treatments, including notably use or re-use of surgery, radiotherapy, hedgehog inhibitors.
   * Non-metastatic cSCC patients:

     * either advanced SCC for which a simple surgical excision is difficult or impossible, or
     * common SCC at high risk of recurrence, for which surgery alone is deemed uncertain by the tumor board, according to EADO /EORTC interdisciplinary guidelines [2]. Patients must either (i) have already received, or (ii) have progressed after, or (iii) be resistant to, or (iv) not be candidate to all possible alternative treatments, including notably use or re-use of surgery, radiotherapy, cetuximab and/or other anti-PD1 checkpoint inhibitors.
   * KA: particularly when surgical excision is considered as too much mutilating for this type of tumor
   * MCC: particularly when either primary tumor is considered unresectable, or skin metastases or local relapse are primarily or secondarily resistant to anti-PD1 (progress under anti-PD1). Patients must either (i) have already received, or (ii) have progressed after, or (iii) be resistant to, or (iv) not be candidate to all possible alternative treatments, including notably use or re-use of surgery, radiotherapy, and/or any anti-PD1 checkpoint inhibitors.
   * CTCL: Tumoral stage of Mycosis fungoides subtypes which are resistant to usual systemic treatments. In order to validate the first inclusion criterion of this trial, the tumor board will take into account that the treatment under investigation is intended to be only a palliative local therapy and cannot compete with a general efficacious strategy, if any.
   * KS: Classic or endemic, histologically confirmed KS, particularly when local response can be considered of either functional or cosmetic benefit. In order to validate the first inclusion criterion of this trial, the tumor board will take into account that the treatment under investigation is intended to be only a palliative local therapy and cannot compete with a general efficacious strategy, if any.
   * MATS: Advanced or refractory MATS.
5. Subjects must have radiographically or clinically measurable disease, defined as at least one injectable lesion that is ≥ 10 mm in diameter in at least 1 dimension, or an aggregate of injectable lesions that measures ≥ 10 mm in diameter in at least 1 dimension.
6. Subjects must be able and willing to undergo serial biopsies of injected lesion(s) and, when applicable and clinically feasible, non-injected lesions.
7. Male or female patients from the age of 18 years.
8. ECOG Performance Status/WHO Performance Status ≤ 1.
9. Hemoglobin > 10.0 g/dL.
10. Platelets > 100 x 109/L.
11. ALT and AST, GGT and Lipase ≤ 1.5 x the upper limit of normal (ULN).
12. Serum creatinine < 1.5 x ULN and GFR > 60 mL/min.
13. All acute toxic effects (excluding alopecia) of any prior therapy must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v. 5.0) Grade ≤ 1 unless otherwise specified.
14. Women of childbearing potential (WOCBP) must have negative pregnancy test results at screening. WOCBP must be using, from screening to three months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomised partner.
15. Male patients with WOCBP partners must agree to use simultaneously two acceptable methods of contraception (i.e. spermicidal gel plus condom) from the screening to three months following the last study drug administration.
16. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Previous or concurrent cancer type that is distinct from the cancers being evaluated in this study, exception made for any other cancer curatively treated ≥ 2 years prior to study entry. Patients suffering from cSCC post-organ transplantation, or cSCC patients with concomitant chronic lymphocytic leukemia are excluded from the study.
2. Previous topical or systemic chemotherapy, immunotherapy, or radiation therapy at the tumor sites within 4 weeks prior to study drug administration.
3. Presence of active severe bacterial or viral infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study. In particular, a documented test for HIV, HBV, HCV and Covid-19 excluding active infection is needed.
4. Impaired cardiocirculatory functions due to any of the following conditions:

   1. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
   2. Inadequately controlled cardiac arrhythmias including atrial fibrillation.
   3. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
   4. Any abnormalities observed during baseline ECG and Echocardiogram investigations that are considered as clinically significant by the investigator.
   5. Uncontrolled hypertension.
   6. Ischemic peripheral vascular disease (Grade IIb-IV).
5. Known arterial aneurysms.
6. INR > 3.
7. Known uncontrolled coagulopathy or bleeding disorder.
8. Known hepatic cirrhosis or severe pre-existing hepatic impairment.
9. Moderate to severe respiratory failure.
10. Active autoimmune disease.
11. Patient requires or is taking systemic corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions and asthma/COPD is not considered an exclusion criterion.
12. Known history of allergy to IL2, TNF, or other human proteins/peptides/antibodies.
13. Pregnancy or breast-feeding.
14. Severe diabetic retinopathy.
15. Recovery from major trauma including surgery within 4 weeks prior to enrollment.
16. Patient with iatrogenic or pathologic severe immune suppression.
17. Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Confirmed best overall response rate (BORR) | Visit will be performed at week 12
  Efficacy of L19IL2/L19TNF measured as Confirmed best overall response rate (BORR) [Complete Response (CR) + Partial Response (PR)] for each tumor type measured according to RECIST v1.1 criteria. Confirmation of CR requires histopathological analysis of exeresis specimens for lesions removed by surgery or of biopsies in all other cases.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Visits will be performed at week 12, week 20, week 28, week 36, week 44 and week 52
  Disease control rate (DCR) [Complete Response (CR) + Partial Response (PR) + Stable Disease (SD)] for each tumor type measured according to RECIST v1.1 criteria.
Local PFS (LPFS) | Visits will be performed at week 12, week 20, week 28, week 36, week 44 and week 52
  Local Progression Free Survival (LPFS) on the treated tumors only
Progression-free survival (PFS) | Visits will be performed at week 12, week 20, week 28, week 36, week 44 and week 52
  Progression-free survival (PFS), assessed separately in patients who are not resected after curative intention and in patients who undergo secondary surgery (neoadjuvant intention), whatever the RECIST response to treatment, taking into account appearance of new lesions and occurrence of metastases,
Adverse Events (AE) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of the trial (week 52).
  Percentage of Patients in Each Treatment Group with AEs, AEs with CTCAE grade ≥3
Serious Adverse Event (SAEs) | From the inclusion in the study (signature of the informed consent form - ICF) until the end of the trial (week 52).
  Percentage of Patients in Each Treatment Group with Drug-Related Adverse Events, Serious Adverse Event (SAEs)
Human anti-fusion protein antibodies (HAFA) | At week 1, at week 4 and at week 12
  Assessment of the formation of human anti-fusion protein antibodies (HAFA) against L19IL2 and L19TNF

CONTACTS AND LOCATIONS:
Locations (14):
- France (3):
  - Hôpital de la Timone, Marseille
  - CHU de Nantes - Hôpital Dieu, Nantes
  - Institut Gustave Roussy, Villejuif
- Italy (8):
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Istituto Nazionale dei Tumori Fondazione IRCCS, Milan
  - IRCCS Istituto Nazionale Tumori "Fondazione Giovanni Pascale", Napoli
  - Istituto Oncologico Veneto IOV, Padua
  - IFO- Istituto Dermatologico San Gallicano, Roma
  - Fondazione Policlinico Universitario A. Gemelli Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliero Universitaria Senese Policlinico Le Scotte, Siena
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), Trieste
- Spain (3):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No